CLINICAL TRIAL: NCT02092077
Title: A Phase 2, Randomized, Open-Label, Safety and Dose-Finding Study Comparing 3 Different Doses of Weekly TV-1106 and Daily Recombinant Human Growth Hormone Therapy in Treatment-Naive, Pre-Pubertal, Growth Hormone-Deficient Children
Brief Title: A Phase 2, Safety and Dose-Finding Study in Treatment-Naive, Pre-Pubertal, Growth Hormone-Deficient Children
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Teva Pharmaceutical Industries, Ltd. (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TV1106-IMM-20001; 2013-004468-69 (EudraCT Number)
Record Dates: First submitted 2014-03-14; First posted 2014-03-19 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Growth Hormone-Deficiency
Keywords: Growth Hormone-Deficient; recombinant human growth hormone
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — albusomatropin; Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- TV-1106 0.554 mg (Experimental)
  Interventions: Drug: TV-1106
- TV-1106 0.924 mg/kg (Experimental)
  Interventions: Drug: TV-1106
- TV-1106 1.20 mg/kg (Experimental)
  Interventions: Drug: TV-1106
- somatropin 0.033 mg/kg/day (Active Comparator): Dosages may be adjusted according to findings and as necessary
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: TV-1106 — TV-1106 0.554mg, TV-1106 0.924 mg, TV-1106 1.20 mg
  Other Names: albutropin; Human Growth Hormone Therapy
  Arms: TV-1106 0.554 mg; TV-1106 0.924 mg/kg; TV-1106 1.20 mg/kg
Drug: somatropin — Dose may be adjusted as required
  Other Names: Human Growth Hormone Therapy
  Arms: somatropin 0.033 mg/kg/day

SUMMARY:
The purpose of this study is to support selection of an appropriate safe and efficacious dose for study in further development.

ELIGIBILITY:
Criteria for Inclusion:

* Pre-pubertal boys ≥ 3 years to ≤ 11 years and pre-pubertal girls ≥ 3 years to ≤ 10 years growth hormone (GH) insufficiency
* Diagnosis criteria consistent with growth hormone research society consensus guidelines
* Patients with a previously treated pituitary tumor must have no tumor progression for at least the past year
* Physician determined rate of change in height less than 2 standard deviations per age group.
* Written Informed Consent
* Parent or legal guardian who is capable and willing to administer the study drug.
* Other criteria apply, please contact the investigator for more information

Criteria for Exclusion:

* Any clinically significant medical condition as determined by the investigator, that is likely to affect growth
* Contraindications to rhGH treatment;
* History of or currently active malignancy, including pituitary tumors;
* Bone age, greater than chronological age or greater than 9 for girls or greater than 10 for boys within 3 months of screening.
* Patients with known diagnosis of diabetes or pre-diabetes
* Growth altering medications
* Allergies to the study medication components;
* Participation in another investigational study within 30 days of screening
* Any medical condition as judged by the investigator to interfere with patient participation or the objectives of the study
* Other criteria apply, please contact the investigator for more information

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2014-04-30 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Height velocity (HV) | Month 6

SECONDARY OUTCOMES:
Height velocity standard deviation score (HV-SDS) | Months 6 and 12
Height standard deviation score (H-SDS) | Months 6 and 12
Number of participants with adverse events | up to 24 months
Height velocity (HV) | Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (34):
- Teva Investigational Site 68016, Minsk, Belarus
- Teva Investigational Site 59060, Varna, Bulgaria
- Georgia (3):
  - Teva Investigational Site 81022, Tbilisi
  - Teva Investigational Site 81023, Tbilisi
  - Teva Investigational Site 81025, Tbilisi
- Teva Investigational Site 63046, Athens, Greece
- Hungary (3):
  - Teva Investigational Site 51159, Budapest
  - Teva Investigational Site 51160, Budapest
  - Teva Investigational Site 51181, Szombathely
- Israel (4):
  - Teva Investigational Site 80052, Afula
  - Teva Investigational Site 80055, Beersheba
  - Teva Investigational Site 80053, Petah Tikva
  - Teva Investigational Site 80056, Ramat Gan
- Teva Investigational Site 53216, Warsaw, Poland
- Teva Investigational Site 52056, Timișoara, Romania
- Russia (10):
  - Teva Investigational Site 50261, Izhevsk
  - Teva Investigational Site 50260, Kazan'
  - Teva Investigational Site 50258, Moscow
  - Teva Investigational Site 50259, Moscow
  - Teva Investigational Site 50264, Novosibirsk
  - Teva Investigational Site 50267, Saint Petersburg
  - Teva Investigational Site 50268, Samara
  - Teva Investigational Site 50263, Saratov
  - Teva Investigational Site 50262, Tomsk
  - Teva Investigational Site 50265, Ufa
- Serbia (2):
  - Teva Investigational Site 61030, Belgrade
  - Teva Investigational Site 61032, Niš
- Teva Investigational Site 31099, Girona, Spain
- Turkey (Türkiye) (2):
  - Teva Investigational Site 82011, Ankara
  - Teva Investigational Site 82013, Aydin
- Ukraine (4):
  - Teva Investigational Site 58138, Kharkiv
  - Teva Investigational Site 58140, Kiev
  - Teva Investigational Site 58139, Kyiv
  - Teva Investigational Site 58142, Odesa